CLINICAL TRIAL: NCT05541835
Title: Hematological Abnormalities In Children With Congenital Cyanotic Heart Disease Attending Assiut University Hospitals: A Prospective Hospital- Based Study.
Brief Title: Hematological Abnormalities in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud abdelshakour, Hematological Abnormalities In Childern With Congenital Cyanotic Heart Disease Attending Assiut University Hospitals: A Prospective Hospital- Based Study, Assiut University
Other Study IDs: Hematological Abnormalities
Record Dates: First submitted 2022-06-25; First posted 2022-09-15 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sampling — venous sampling of patient

SUMMARY:
the aim of the study is to determine Hematological abnormalities in Congenital Cyanotic Heart Disease

DETAILED DESCRIPTION:
Congenital heart defects are the most common developmental anomaly and are the commonest noninfectious causes of mortality in newborns; they affect up 1000 infants and in most cases the cause is unknown . Erythrocytosis, thrombocytopenia, platelets function defects, coagulation factors deficiencies are the main hematologic disorders in patients with cyanotic congenital heart disease .The hemorrhagic tendency was initially attributed to an increase in tissue vascularity, but co-existing hemostatic defects were subsequently identified and attributed to thrombocytopenia, shortened platelet survival, and deficient von Willebrand multimers .

In patients , platelets are shown to have both qualitative and quantitative abnormalities.However, there are conflicting data as regards the etiology of thrombocytopenia in congenital cyanotic heart disease . significant association has been reported between thrombocytopenia and a high hematocrit in cyanotic patients and multiple etiologies has been suggested including chronic compensated disseminated intravascular coagulation (DIC), reduce synthesis of clot factors and/or deranged platelet aggregation. Immature reticulated platelets represent the youngest platelets released into the circulation by regenerated marrow megakaryocyte and are the analogue of the red cell reticulocyte .The rate of platelet turnover can be evaluated by the relationship between the percent of reticulated platelets and the platelet count.

Erythrocytosis is an isolated increase in the number of red blood cells. Primary erythrocytosis is an increased red cell mass which surfaces in the absence of a definable stimulus, whereas secondary erythrocytosis refers to an isolated increase in the red cell mass in response to such stimulus as low systemic arterial oxygen saturation in the context of cyanotic congenital heart disease. Polycythemia could often be beneficial. Yet, it poses certain risks to the microcirculation. This is mainly because the capillary diameter is significantly smaller than the red cell diameter and this mismatch could cause viscosity

To increase at the capillary level. Patients with cyanotic heart disease may have an acceptable quality of life. However, they are invariably prone to several complications. For instance, hyperviscosity, hyperuricemia (mainly due to age-related impairment of uric acid excretion in adults), thrombocytopenia (decreased level of platelet production), blood clotting abnormalities (reduced synthesis of clotting factors and/or deranged platelet aggregation), cerebral abscess, cerebral embolism and endocarditis .

ELIGIBILITY:
Inclusion Criteria:

* All children.
* congenital cyanotic heart disease

Exclusion Criteria:

* other congenital heart disease.
* other congenital anomalies.
* other chronic disease.
* post-operative patient.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All childern with Cyanotic Congenital heart disease admitted to the pediatric cardiology unit of Assiut University Hospitals over a period of one year
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Hematological Abnormalities In ChilCongenital congenital Cyanotic Heart Disease | Baseline
  Determine hematological abnormality

SECONDARY OUTCOMES:
Children with Congenital Cyanotic Heart Disease | Baseline
  To change morbidity and mortality, number of death in children with congenital cyanotic heart disease.